CLINICAL TRIAL: NCT03563144
Title: QUILT-3.088 NANT Pancreatic Cancer Vaccine: Phase II Randomized Trial of the NANT Pancreatic Cancer Vaccine vs. Standard-of-Care as First- Line Treatment for Patients With Metastatic Pancreatic Cancer
Brief Title: QUILT-3.088: NANT Pancreatic Cancer Vaccine
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Trial not initiated
Sponsor: ImmunityBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QUILT-3.088
Record Dates: First submitted 2018-05-25; First posted 2018-06-20 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2018-08

CONDITIONS: Metastatic Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; 130-nm albumin-bound paclitaxel; ALT-803; yeast-CEA vaccine; avelumab; Bevacizumab; Capecitabine; Cyclophosphamide; Fluorouracil; Leucovorin; Oxaliplatin

STUDY DESIGN:
Intervention Model Description: This is a randomized parallel group study comparing the NANT Pancreatic Cancer Vaccine and standard therapy with respect to efficacy and safety in treatment naïve patients with pancreatic cancer. Patients will be stratified by ECOG status and then randomized 1:1 to receive either the NANT Pancreatic Vaccine (n~532) or standard therapy with gemcitabine alone (ECOG 2; n~266) or combined with nab-paclitaxel (ECOG 0-1; n~266). Treatment may continue for up to 2 years or until documented progression (RECIST v 1.1) or unacceptable toxicity. Patients on standard therapy who progress or experience unacceptable toxicity may crossover to receive NANT Pancreatic Vaccine.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- NANT Pancreatic Cancer Vaccine (Experimental): in subjects with ECOG=2 or subjects with ECOG=0 or 1
  A combination of agents will be administered to subjects in this study:
  cyclophosphamide, bevacizumab, oxaliplatin, capecitabine, 5-fluorouracil, leucovorin, nab-paclitaxel, aldoxorubicin HCl, avelumab, ALT-803, haNK, GI-4000, GI-6207, GI-6301, ETBX-011, ETBX-021, ETBX-051, ETBX-061.
  Interventions: Drug: Nab-paclitaxel; Drug: Aldoxorubicin HCl; Biological: ALT-803; Biological: ETBX-011; Biological: ETBX-021; Biological: ETBX-051; Biological: ETBX-061; Biological: GI-4000; Biological: GI-6207; Biological: GI-6301; Biological: haNK; Drug: Avelumab; Drug: Bevacizumab; Drug: Capecitabine; Drug: Cyclophosphamide; Drug: 5-Fluorouracil; Drug: Leucovorin; Drug: Oxaliplatin
- Gemcitabine and Nab-paclitaxel (Active Comparator): Gemcitabine plus Nab-paclitaxel will be administered to subjects with ECOG=2
  Interventions: Drug: Gemcitabine; Drug: Nab-paclitaxel
- Gemcitabine (Active Comparator): Gemcitabine will be administered to subjects with ECOG=0 or 1
  Interventions: Drug: Gemcitabine

INTERVENTIONS:
Drug: Gemcitabine — Gemcitabine is a type of chemotherapy medication used to interfere with the cancer cells' ability to grow and divide.
  Arms: Gemcitabine; Gemcitabine and Nab-paclitaxel
Drug: Nab-paclitaxel — NAB-paclitaxel is a type of chemotherapy called a microtubule inhibitor. Microtubule inhibitors interfere with a cancer cell's ability to grow and divide.
  Arms: Gemcitabine and Nab-paclitaxel; NANT Pancreatic Cancer Vaccine
Drug: Aldoxorubicin HCl — Albumin-binding prodrug of doxorubicin HCl
  Arms: NANT Pancreatic Cancer Vaccine
Biological: ALT-803 — Recombinant human super agonist interleukin-15 (IL-15) complex
  Arms: NANT Pancreatic Cancer Vaccine
Biological: ETBX-011 — Ad5 [E1-, E2b-]-CEA
  Arms: NANT Pancreatic Cancer Vaccine
Biological: ETBX-021 — Ad5 [E1-, E2b-]-human epidermal growth factor receptor 2 [HER2] vaccine
  Arms: NANT Pancreatic Cancer Vaccine
Biological: ETBX-051 — Ad5 [E1-, E2b-]-Brachyury vaccine
  Arms: NANT Pancreatic Cancer Vaccine
Biological: ETBX-061 — Ad5 [E1-, E2b-]-mucin 1[MUC1]
  Arms: NANT Pancreatic Cancer Vaccine
Biological: GI-4000 — Vaccine derived from recombinant Saccharomyces cerevisiae yeast expressing mutant Ras proteins
  Arms: NANT Pancreatic Cancer Vaccine
Biological: GI-6207 — CEA yeast vaccine
  Arms: NANT Pancreatic Cancer Vaccine
Biological: GI-6301 — Brachyury yeast vaccine
  Arms: NANT Pancreatic Cancer Vaccine
Biological: haNK — NK-92 [CD16.158V, ER IL-2]
  Arms: NANT Pancreatic Cancer Vaccine
Drug: Avelumab — Avelumab
  Arms: NANT Pancreatic Cancer Vaccine
Drug: Bevacizumab — Bevacizumab
  Arms: NANT Pancreatic Cancer Vaccine
Drug: Capecitabine — Capecitabine
  Arms: NANT Pancreatic Cancer Vaccine
Drug: Cyclophosphamide — 2-[bis(2-chloroethyl)amino]tetrahydro-2H-1,3,2-oxazaphosphorine 2-oxide monohydrate
  Arms: NANT Pancreatic Cancer Vaccine
Drug: 5-Fluorouracil — 5-fluoro-2,4 (1H,3H)-pyrimidinedione
  Arms: NANT Pancreatic Cancer Vaccine
Drug: Leucovorin — L-Glutamic acid, N-[4-[[(2-amino-5-formyl-1,4,5,6,7,8-hexahydro-4-oxo-6-pteridinyl)methyl]amino]benzoyl]-, calcium salt
  Arms: NANT Pancreatic Cancer Vaccine
Drug: Oxaliplatin — Oxaliplatin
  Arms: NANT Pancreatic Cancer Vaccine

SUMMARY:
QUILT-3.088 NANT Pancreatic Cancer Vaccine: Phase II Randomized Trial of the NANT Pancreatic Cancer Vaccine vs. Standard-of-Care as First- Line Treatment for Patients with Metastatic Pancreatic Cancer.

DETAILED DESCRIPTION:
This is a two-cohort, open-label, randomized phase 2 study to evaluate the safety and efficacy (as assessed by PFS) of the NANT Pancreatic Cancer Vaccine regimen (experimental arms) vs SoC therapy (control arms) as first-line treatment for subjects with metastatic pancreatic cancer.

Subjects will be enrolled into two independent cohorts based on ECOG status. Subjects with ECOG 0-1 will be randomized 1:1 to receive the NANT Pancreatic Cancer Vaccine regimen (experimental arm) or gemcitabine in combination with nab-paclitaxel (control arm), while subjects with ECOG 2 will be randomized 1:1 to receive the NANT Pancreatic Cancer Vaccine regimen (experimental arm) or gemcitabine monotherapy (control arm).

The experimental arms will be administered in two phases, an induction and a subsequent maintenance phase. The treatment regimen administered in the experimental arms will be identical for all subjects, independent of ECOG status. Subjects may continue induction treatment for up to 1 year. Those who have a complete response (CR) in the induction phase will enter the maintenance phase of the study. Subjects who experience ongoing stable disease (SD) or an ongoing partial response (PR) after 1 year of induction phase treatment may enter the maintenance phase at the Investigator's discretion. Subjects may remain on the maintenance phase of the study for up to 1 year.

Treatment in the study will be discontinued if the subject experiences confirmed PD or unacceptable toxicity, withdraws consent, or if the Investigator feels it is no longer in the subject's best interest to continue treatment. Subjects receiving treatment in the control arms may cross over to treatment in the induction phase of the experimental arms after experiencing PD. Subjects receiving treatment in the experimental arms with an initial assessment of PD per RECIST 1.1 may, at the discretion of the Investigator, continue to receive study treatment until PD is confirmed. The maximum time on study treatment is 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old.
2. Able to understand and provide a signed informed consent that fulfills the relevant IRB or Independent Ethics Committee (IEC) guidelines.
3. Histologically-confirmed metastatic pancreatic adenocarcinoma that has not been previously treated with chemotherapy.
4. ECOG performance status of 0-2.
5. Have at least 1 measurable lesion of ≥ 1.0 cm.
6. If available, must be willing to release a recent formalin-fixed, paraffin-embedded (FFPE) tumor biopsy specimen for prospective and exploratory tumor molecular profiling. If an historic specimen is not available, the subject must be willing to undergo a biopsy during the screening period, if considered safe by the Investigator.
7. Must be willing to provide blood samples prior to the start of treatment on this study for prospective tumor molecular profiling and exploratory analyses.
8. Must be willing to provide a tumor biopsy specimen 8 weeks after the start of treatment for exploratory analyses, if considered safe by the Investigator.
9. Ability to attend required study visits and return for adequate follow-up, as required by this protocol.
10. Agreement to practice effective contraception for female subjects of child-bearing potential and non-sterile males. Female subjects of child-bearing potential must agree to use effective contraception for up to 1 year after completion of therapy, and non-sterile male subjects must agree to use a condom for up to 4 months after treatment. Effective contraception includes surgical sterilization (eg, vasectomy, tubal ligation), two forms of barrier methods (eg, condom, diaphragm) used with spermicide, intrauterine devices (IUDs), and abstinence.

Exclusion Criteria:

1. Serious uncontrolled concomitant disease that would contraindicate the use of the investigational drug used in this study or that would put the subject at high risk for treatment-related complications.
2. Systemic autoimmune disease (eg, lupus erythematosus, rheumatoid arthritis, Addison's disease, autoimmune disease associated with lymphoma).
3. History of organ transplant requiring immunosuppression.
4. History of or active inflammatory bowel disease (eg, Crohn's disease, ulcerative colitis).
5. Inadequate organ function, evidenced by the following laboratory results:

   1. Absolute neutrophil count (ANC) < 1,000 cells/mm^3.
   2. Platelet count < 75,000 cells/mm^3.
   3. Total bilirubin greater than the upper limit of normal (ULN; unless the subject has documented Gilbert's syndrome).
   4. Aspartate aminotransferase (AST [SGOT]) or alanine aminotransferase (ALT [SGPT]) > 2.5 × ULN (> 5 × ULN in subjects with liver metastases).
   5. Alkaline phosphatase levels (ALP) > 2.5 × ULN (> 5 × ULN in subjects with liver metastases, or >10 × ULN in subjects with bone metastases).
   6. Serum creatinine > 2.0 mg/dL or 177 μmol/L.
   7. Serum anion gap > 16 mEq/L or arterial blood with pH < 7.3.
   8. Medically uncorrectable grade 3 anemia (hemoglobin < 8 g/dL).
6. Uncontrolled hypertension (systolic > 160 mm Hg and/or diastolic > 110 mm Hg) or clinically significant (ie, active) cardiovascular disease, cerebrovascular accident/stroke, or myocardial infarction within 6 months prior to first study medication; unstable angina; congestive heart failure of New York Heart Association grade 2 or higher; or serious cardiac arrhythmia requiring medication. Subjects with uncontrolled hypertension should be medically managed on a stable regimen to control hypertension prior to study entry.
7. Serious myocardial dysfunction defined by echocardiogram (ECHO) as absolute left ventricular ejection fraction (LVEF) 10% below the institution's lower limit of predicted normal.
8. Dyspnea at rest due to complications of advanced malignancy or other disease requiring continuous oxygen therapy.
9. Positive results of screening test for human immunodeficiency virus (HIV).
10. Current chronic daily treatment (continuous for > 3 months) with systemic corticosteroids (dose equivalent to or greater than 10 mg/day methylprednisolone), excluding inhaled steroids. Short-term steroid use to prevent IV contrast allergic reaction or anaphylaxis in subjects who have known contrast allergies is allowed.
11. Known hypersensitivity to any component of the study medication(s).
12. Subjects taking any medication(s) (herbal or prescribed) known to have an adverse drug reaction with any of the study medications.
13. Concurrent or prior use of a strong cytochrome P450 (CYP)3A4 inhibitor (including ketoconazole, itraconazole, posaconazole, clarithromycin, indinavir, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, voriconazole, and grapefruit products) or strong CYP3A4 inducers (including phenytoin, carbamazepine, rifampin, rifabutin, rifapentin, phenobarbital, and St John's Wort) within 14 days before study day 1.
14. Concurrent or prior use of a strong CYP2C8 inhibitor (gemfibrozil) or moderate CYP2C8 inducer (rifampin) within 14 days before study day 1.
15. History of receiving any investigational treatment for metastatic pancreatic cancer, or participation in an investigational drug study within 30 days prior to screening for this study, except for testosterone-lowering therapy in men with prostate cancer.
16. Assessed by the Investigator to be unable or unwilling to comply with the requirements of the protocol.
17. Concurrent participation in any interventional clinical trial.
18. Pregnant and nursing women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-08 (Estimated); Primary Completion 2019-12-30 (Estimated); Study Completion 2022-02-09 (Actual)

PRIMARY OUTCOMES:
Progression-Free Survival | 12 mths
  Compare the efficacy of the NANT Pancreatic Cancer Vaccine regimen vs standard-of-care (SoC) therapy as first-line treatment for patients with metastatic pancreatic cancer as assessed by progression-free survival (PFS) using RECIST Version 1.1

SECONDARY OUTCOMES:
Overall Survival | 24 months
  Overall Survival from first treatment to date of death (any cause)
Overall Response Rate | 19 months
  Overall Response Rate, as determined by the percentage of patients achieving Partial or Complete response per RECIST 1.1 and irRC
Duration of Response | 19 months
  Duration of Response from date of first response to date of disease progression or death (any cause), per RECIST 1.1 and irRC
Disease Control Rate | 19 months
  Disease Control Rate: the number of patients with a CR, PR or SD lasting at least 2 months per RECIST 1.1 and irRC
Quality of Life by Patient-Reported Outcomes | 19 months
  Quality of Life as assessed by Patient Reported Outcomes using the FACT-C questionnaire
Progression Free Survival | 12 months
  Progression Free Survival from baseline to progression per irRC
Evaluation of safety as determined by incidence or treatment-emergent adverse events | 19 months
  Incidence of treatment -emergent adverse events using NCI CTCAE Version 4.03

CONTACTS AND LOCATIONS:
Locations (1):
- Chan Soon-Shiong Institute for Medicine, El Segundo, California, United States

IPD SHARING:
Plan to Share IPD: Undecided